CLINICAL TRIAL: NCT01799538
Title: Bronchodilator Effects of Nebulized Versus Inhaled Albuterol in Subjects With Lymphangioleiomyomatosis
Brief Title: Nebulized or Inhaled Albuterol for Lymphangioleiomyomatosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130051; 13-H-0051
Record Dates: First submitted 2013-02-23; First posted 2013-02-26 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-04-04

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Albuterol; Bronchodilator; Nebulizer; Metered Dose Inhaler
MeSH Terms: conditions — Lymphangioleiomyomatosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Nebullizer
  Interventions: Drug: albuterol nebulizer; Procedure: PFT
- 2 (Active Comparator): Inhaler
  Interventions: Drug: albuterol inhaler; Procedure: PFT

INTERVENTIONS:
Drug: albuterol inhaler — 2 puffs of Metered Dose inhaler for Bronchodilation
  Arms: 2
Drug: albuterol nebulizer — Albuterol administered by nebulization will produce a greater increase in FEV1
  Arms: 1
Procedure: PFT — Breathing Test

SUMMARY:
Background:

- Lymphangioleiomyomatosis (LAM) is a rare type of lung disease that occurs almost exclusively in women. In LAM, muscle tissue grows in the lungs and starts to block the flow of air. It is a progressive disease, and in severe cases may require a lung transplant. One possible treatment to improve breathing in people with LAM is inhaled albuterol. Albuterol can be given in a metered dose inhaler (MDI) or with a nebulizer. Researchers want to compare these methods to see which method best improves lung function in women with LAM.

Objectives:

- To see whether a nebulizer or MDI can better improve lung function in women with LAM.

Eligibility:

- Women at least 18 years of age who have impaired lung function because of LAM.

Design:

* Participants will be screened with a physical exam and medical history. No lab tests will be needed for this study.
* Participants will have a 3-day overnight stay at the National Institutes of Health. Those who are using long-acting inhalers will have to stop taking these drugs 1 week before the study.
* Participants will receive either the nebulizer or two or four puffs of the inhaler. Four puffs of albuterol is a higher dose than is normally prescribed, and is being tested on this study.
* Participants will have each treatment around the same time of day on each of the 3 days. Before and after taking the albuterol, participants will have lung function tests.

DETAILED DESCRIPTION:
We have reported that approximately one third of patients with lymphangioleiomyomatosis (LAM) who have airflow obstruction respond to bronchodilators such as albuterol, a Beta2-adenergic receptor agonist, with an increase in forced expiratory flow in one second (FEV1) of 12% and 200 ml above baseline values. Others however, have questioned these findings, reporting instead, a low rate of response of only six percent. Contrasting with our study, in this study albuterol was administered with a metered dose inhaler whereas in ours it was given by nebulizer. We propose to measure changes in lung function after administration of albuterol, respectively by metered inhaler and nebulizer, for 3 consecutive days in 100 LAM subjects. Our hypothesis is that albuterol administered by nebulization will produce a greater increase in FEV1 than two puffs of inhaled albuterol. If this hypothesis is confirmed, then we may recommend that patients with LAM and airflow obstruction use as a method of drug administration a nebulizer, rather than a metered dose inhaler.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of LAM either by tissue biopsy, evidence of lung and other organ involvement (renal angiomyolipomas, chylous effusions, lymphangioleiomyomas), high serum levels of vascular endothelial growth factor D (VGEF-D)(1) or a diagnosis of TSC associated with cystic lung lesions.
* Age 18 years or over
* Evidence of airflow obstruction: FEV1/VC ratio < fifth percentile of predicted normal and an FEV(1) <80% predicted of the normal values.

EXCLUSION CRITERIA:

Subjects will be excluded from the study if they meet one or more of the following criteria:

* History of hypersensitivity to albuterol or any of its components.
* Moderate or large pleural effusions (chest x-ray and or CT scan procedure completed under Protocol 95-H-0186)
* History of seizures other than during infancy
* Inability to withhold bronchodilators for 24 hours
* Cognitive Impairment
* Age less than 18 years
* Male sex
* Status-post lung or kidney transplantation
* Pregnant or breast feeding (women of childbearing potential will undergo a blood or urine pregnancy test under Protocol 95-H-0186).
* Treatment with monoaminoxidase inhibitors, tricyclic antidepressants or Beta-adrenergic receptor antagonists or long acting anticholinergic bronchodilators who are unable to be discontinued for at least seven days before enrollment.
* Patients with URI, uncontrolled hyperthyroidism or severe gastro-esophageal reflux. Major systemic diseases (i.e., malignancy; myocardial infarction or unstable angina; type 1 diabetes, severe hypertension; liver cirrhosis).

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06-10 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Greater improvement in lung function with nebulized albuterol. | 3 days
  Greater improvement in lung function with nebulized albuterol.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCormack FX. Lymphangioleiomyomatosis: a clinical update. Chest. 2008 Feb;133(2):507-16. doi: 10.1378/chest.07-0898. PMID 18252917
- [Background] Ryu JH, Moss J, Beck GJ, Lee JC, Brown KK, Chapman JT, Finlay GA, Olson EJ, Ruoss SJ, Maurer JR, Raffin TA, Peavy HH, McCarthy K, Taveira-Dasilva A, McCormack FX, Avila NA, Decastro RM, Jacobs SS, Stylianou M, Fanburg BL; NHLBI LAM Registry Group. The NHLBI lymphangioleiomyomatosis registry: characteristics of 230 patients at enrollment. Am J Respir Crit Care Med. 2006 Jan 1;173(1):105-11. doi: 10.1164/rccm.200409-1298OC. Epub 2005 Oct 6. PMID 16210669
- [Background] Costello LC, Hartman TE, Ryu JH. High frequency of pulmonary lymphangioleiomyomatosis in women with tuberous sclerosis complex. Mayo Clin Proc. 2000 Jun;75(6):591-4. doi: 10.4065/75.6.591. PMID 10852420
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-H-0051.html